CLINICAL TRIAL: NCT05356936
Title: Pilot Study of Vitamin K2 (MK-7) and Vitamin D3 Supplementation and the Effects on PASC Symptomatology and Inflammatory Biomarkers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Grace McComsey, Vice President of Research, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY20220109
Record Dates: First submitted 2022-04-26; First posted 2022-05-02 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Post-acute COVID-19 Syndrome
Keywords: Vitamin K2 (MK-7) supplementation; Vitamin D3 supplementation; Inflammatory biomarkers
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome | interventions — Vitamin K 2; Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin K2(MK-7) and Vitamin D3 (Experimental): Participants randomized to this group will receive Vitamin K2 (MK-7) and Vitamin D3 by mouth.
  Interventions: Dietary Supplement: Vitamin K2 (MK-7); Dietary Supplement: Vitamin D3
- Control (No Intervention): Participants to this group will receive no intervention.

INTERVENTIONS:
Dietary Supplement: Vitamin K2 (MK-7) — Participants will receive Vitamin K2 (MK-7) daily by mouth.
  Arms: Vitamin K2(MK-7) and Vitamin D3
Dietary Supplement: Vitamin D3 — Participants will receive Vitamin D3 daily by mouth.
  Arms: Vitamin K2(MK-7) and Vitamin D3

SUMMARY:
Participants are being asked to take part in this research study because they have had a previous diagnosis (at least 3 months ago) of COVID-19 and are experiencing persistent, recurrent or even new symptoms, i.e. post-acute sequelae of SARS-CoV-2 (PASC). The Investigators are interested in studying the effects of Vitamin K2 (MK-7) and Vitamin D3 supplementation on PASC symptoms and the underlying inflammatory process.

ELIGIBILITY:
Inclusion Criteria:

* Previous COVID-19 infection as documented by a positive Nucleic Acid Amplification Test (NAAT) PCR test or any licensed SARS-CoV-2 antigen test kit and prolonged, recurrent or newly developed symptoms more than 3 months after the positive test result.
* Male or Female age ≥18 years
* Provides written informed consent and is capable of reading and comprehending the informed consent
* Able to swallow pills.
* No active nausea, vomiting
* All women of child-bearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 72 hours prior to start of study medication. WOCBP is defined as any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy), who is not postmenopausal (defined as amenorrhea for 12 consecutive months), or is on hormone replacement therapy (HRT) with documented plasma follicle-stimulating hormone level 35mLU/mL. Women who are using oral, implanted, or injectable contraceptive hormones or mechanical products such as an intrauterine device or barrier methods (diaphragm, condoms, spermicides) to prevent pregnancy or practicing abstinence or where partner is sterile (e.g., vasectomy), should be considered to be of child bearing potential.
* Female subjects who are not of reproductive potential (have reached menopause or undergone hysterectomy, bilateral oophorectomy or tubal ligation) or whose male partner has undergone successful vasectomy with resulting azoospermia or has azoospermia for any other reason, are eligible without requiring the use of contraception. Acceptable documentation of menopause, sterilization, and azoospermia is patient reported history.
* All subjects must not participate in a conception process (e.g. active attempt to become pregnant or to impregnate, sperm donation, in vitro fertilization), and if participating in sexual activity that could lead to pregnancy, the female subject/male partner must use condoms (male or female) in addition to one of the following forms of contraception while on study: either a spermicidal agent, diaphragm, cervical cap, IUD, or hormonal-based contraception.

Exclusion Criteria:

* Subjects unable to consent due to language barrier or cognitive impairment.
* Pregnancy/lactation.
* Regular use of agents that may affect inflammation in the last 3 months. The regular use of NSAIDS, aspirin, or statins will be allowed as long as dose has been stable for the last 3 months and is not expected to change during the study.
* Subject receiving vitamin K antagonists (e.g. warfarin, coumadin)
* Subject consuming supplements of vitamin K1, K2, or Vitamin D. A daily multivitamin will not be exclusionary as long as vitamin D is not > 600 UI daily.
* Presence of active neoplastic diseases requiring chemotherapy and/or use of immunosuppressive drugs
* BMI <18 kg/m2.
* Allergy or intolerance to vitamin K2 or vitamin D3
* Hospitalization within the previous 28 days.
* Inability or unwillingness of the individual to give written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Change in high-sensitivity C-reactive protein (hs-CRP) as measured by blood test | Baseline, week 12, week 24
Change in interleukin 6 (IL-6) as measured by blood test | Baseline, week 12, week 24
Change in intestinal fatty acid binding protein (Ifab) as measured by blood test | Baseline, week 12, week 24
Change in soluble Tumor Necrosis Factor Receptor II ( sTNF-RII) as measured by blood test | Baseline, week 12, week 24
Change in Vitamin K2 (MK-7) levels as measured by blood test | Baseline, week 12, week 24
Change in Vitamin D3 levels as measured by blood test | Baseline, week 12, week 24

SECONDARY OUTCOMES:
Percent of subjects with >Grade 2 adverse events as measured by patient report | Up to 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Grace McComsey, MD, FIDSA, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No